CLINICAL TRIAL: NCT00386594
Title: Pilot Study of Oral 852A for Elimination of High-Grade Dysplasia in Barrett's Esophagus
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Rogers, B.H. Gerald, M.D. (Individual)
Collaborators: 3M (Industry)
Responsible Party: B. H. Gerald Rogers, M.D., Weiss Memorial Hospital, Chicago, Illinois
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 100606
Record Dates: First submitted 2006-10-08; First posted 2006-10-11 (Estimated); Last update posted 2009-01-21 (Estimated); Status verified 2006-12

CONDITIONS: Barrett Esophagus
Keywords: Barrett Esophagus; High grade dysplasia; Carcinoma in situ; 825A
MeSH Terms: conditions — Barrett Esophagus; Carcinoma in Situ

INTERVENTIONS:
Drug: 852A

SUMMARY:
Barrett's esophagus with high-grade dysplasia is a premalignant condition caused by chronic reflux of gastric contents into the esophagus. High-grade dysplasia is the same as carcinoma-in-situ. If untreated, patients with this condition are at high risk for developing cancer of the esophagus. Cancer of the esophagus is a miserable disease that is difficult to treat and about 95% fatal after 5 years. To prevent progession to cancer of the esophagus several interventions are available and they include surgery, Photofrin photodynamic therapy, endoscopic mucosal resection and endoscopic thermal therapy. All of these modalities are uncomfortable, expensive and have associated risks. The oral agent, 852A stimulates the innate immune system in such a way as to eliminate early cancer. A similar dermatologic drug(imiquimod) is approved for treating the premalignant condition, actinic keratosis. If local therapy with imiquimod can eliminate a premalignant lesion in the skin, a similar acting drug should be able to do the same for a premalignant lesion in the lining of the esophagus. This study is designed to test that hypothesis.

DETAILED DESCRIPTION:
This study is to determine if a locally applied immune response modifier will eliminate high grade dysplasia in Barrett's esophagus. Barrett's esophagus is a premalignant condition caused by chronic reflux of gastric contents into the lower esophagus. Present practice is to do a periodic esophagoscopy on patients with Barrett's esophagus and take biopsies in search of dysplasia. If the pathologist reports low grade dysplasia, the patient usually receives more intensive surveillance. If the pathologist reports high grade dysplasia, the patient and his physician are faced with a dilema. High grade dysplasia is carcinoma in situ and there is a strong propensity for such patients to progess to frank carcinoma of the esophagus. Carcinoma of the esophagus is a miserable disease which is difficult to treat and leads to death in about 95% of the cases at 5 years. The present standard for patients with high grade dysplasia is to recommend esophagectomy. Esophagectomy is a major surgical procedure with significant associated morbidity and mortality. Porfimer sodium(Photofrin) photodynamic therapy is effective in eliminating high grade dysplasia in Barrett's esophagus. It has been approved by the FDA but it is not widely utilized because of its complexity and expense. Other modalities such as endoscopic mucosal resection and endoscopic thermal ablation techiques are being studied. Although endoscopic techniques are much safer than surgery, they all are uncomfortable and carry some risk. Many patients with Barrett's esophagus are elderly and most with high grade dysplasia do not live long enough to develop cancer. This fact has made some gastroenterolgists recommend intensive surveillance as an alternative to the above mentioned therapeutic modalities. Intensive surveillance in this setting means endoscopy with biopsies every 3 months with specific therapy recommended only if frank cancer is found. This study is based upon the fact that intensive surveillance is an acceptable way of following these patients. The only difference is an oral agent will be added in hopes of getting rid of high grade dysplasia. If high grade dysplasia could be eliminated by an oral medication it would be a quantum improvement over what we have. The present belief is if high grade dysplasia is eliminated there would be no progression to cancer.

852A is an immune response modifier being developed by 3M Pharmaceuticals. It is thought to exert its therapeutic effect by simulating alpha interferon. 852A is similar to the immune response modifier imiquimod(Aldara). Imiquimod is presently approved by the precancerous dermatological condition, actinic keratosis. It is very effective. Treatment is simply applying 5% imiquimod cream twice weekly to the skin lesion for 16 weeks. It seems reasonable that if an immune response modifier will eliminate precancerous lesions of the skin by local application, the same should be true for precancerous lesions of the esophagus. In this study 852A will be swallowed to see whether it can eliminate high grade dysplasia from the esophagus.

Entrance into the present study would be predicated on the confirmation of high grade dysplasia in Barrett's esophagus. If the prospective subject meets all of the inclusion and exclusion criteria set out in the protocol, endoscopic ultrasound of the esophagus would be done. If endoscopic ultrasound shows no invasion into the submucosa the patient would be asked to sign an informed consent. Once entered into the sudy the subject would be given the study drug twice weekly, 3-4 days apart, for 8 weeks. 852A will be supplied in sterile vials by 3M Pharmaceuticals. Five mg of 852A will be mixed with sterile 5% dextrose in water to give a final volume of 30 ml. The patient will promply swallow the study drug after it is mixed. The subject will then assume a recumbent position for 30 minutes in hopes that the medication will stay in contact with the mucosa of the esophagus long enough to get an effect. All doses of the study medication will be given in the principal investigator's clinic. After the first dose is given that patient will stay in the clinic under observation for 4 hours. Observation includes taking the temperature, pulse, and blood pressure every hour. If there are no adverse effects after the first dose, the observation period after subsequent doses will reduced to one hour. Laboratory tests will be repeated 1,2,4 and 8 weeks after the first dose is given. As set out in the study protocol, if the patient has any significant adverse event or laboratory deviation, the subject would be dropped from the study. Throughout the study the subjects will be treated with a double dose of a proton pump inhibitor to control gastric acid reflux.

After 8 weeks of therapy the study medication will be stopped. Four weeks thereafter and 12 weeks from the beginning, repeat endosocpy with biopsies will be done. If biopsies show no residual high grade dysplasia, the patient will be continued in an intensive surveillance program. Intensive surveillance means endoscopy with biopsies every 3 months for 1 year, then every 6 months for 1 year then yearly for 3 more years. If high grade dysplsia persists after 8 weeks of treatment or cancer is found, the patient would be referred for conventional therapy. Likewise, if high grade dysplsia recurs or cancer is found during the intensive surveillance program, the subject will be referred for conventional therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, 18 years or older
2. Documented Barrett's esophagus with high-grade dysplasia with diagnosis confirmed by the Pathology Department at the University of Chicago
3. Laboratory parameters within the range given in the protocol.

Exclusion criteria.

1. Patients with high-grade dysplasia of the esophagus who on ultrasound of the esophagus have invasion through the muscularis mucosa
2. Patients who do not tolerate repeated endoscopy
3. Patients who are allergic to 852A or any component in its vehicle
4. Patients with autoimmune disease such as rheumatoid arthritis, ulcerative colitis or Crohn's disease which could be worsened by stimulating the innate immune system
5. Pregnant patients, and vulnerable patients who cannot or will not use contraceptives
6. Males who have a sexual partner who is pregnant or a vulnerable partner who cannot or will not use contraceptives.
7. Cardiac ischemia, cardiac arrhythmias or congestive heart failure uncontrolled by medication
8. History of, or clinical evidence of, a condition which, in the opinion of the investigator, could confound the results of the study or put the subject at undue risk
9. Uncontrolled intercurrent or chronic illness
10. Active hepatitis B or C with evidence of ongoing viral replication
11. Hyperthyroidism
12. Uncontrolled seizure disorder
13. Active coagulation disorder not controlled with medication
14. HIV positive
15. Congenital long QT syndrome or abnormal baseline QTc interval after Bazett's correction
16. Laboratory values outside of the acceptable range as given in protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2006-10; Primary Completion 2010-10 (Estimated); Study Completion 2012-10 (Estimated)

PRIMARY OUTCOMES:
Elimination of high-grade dysplasia in Barrett's esophagus | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: B. H. Gerald Rogers, M. D., Principal Investigator — Clinical Professor, University of Chicago School of Medicine. Attending Physician, Weiss Memorial Hospital, Chicago, Illinois
Locations (2):
- United States (2):
  - B. H. Gerald Rogers, M. D., Chicago, Illinois
  - Weiss Memorial Hospital, Chicago, Illinois